CLINICAL TRIAL: NCT05332197
Title: Yellow Fever Vaccine Booster Trial in Children- a Phase 3 Clinical Trial to Establish Safety and Immunogenicity of Repeated YF Vaccination in Healthy Gambian Children of Different Ages
Brief Title: Booster Vaccine for Yellow Fever
Acronym: BoVY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LEO 26467
Record Dates: First submitted 2022-03-31; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Yellow Fever
Keywords: immunogenicity; Yellow fever vaccine
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 17D Yellow fever vaccine (Experimental): All children will receive a single shot of the 17D Yellow fever vaccine. This vaccine contains the Rockefeller17D-substrain 204 strain of Yellow fever virus. This vaccine is presented as a 10 dose vial with freeze-dried content which is reconstituted with a diluent, provided with the vaccine by the manufacturer. Reconstituted vaccines have to be kept in a vaccine carrier at 2-8°C as per WHO and manufacturer requirements. Any remaining reconstituted vaccine not used has to be discarded after 6 h. The standard dose is 0·5 ml and is administered subcutaneously in the deltoid region using standard vaccination syringes (needle size 25G × 3/4") with a 45° injection angle
  Interventions: Biological: 17D Yellow fever vaccine

INTERVENTIONS:
Biological: 17D Yellow fever vaccine — This vaccine contains the Rockefeller17D-substrain 204 strain of Yellow fever virus. The exact potency of each batch is released with the certificate of analysis that accompanies each batch and the potency confirmed at time of release closest to internal minimum specification. This vaccine is the same vaccine used by the national EPI program

SUMMARY:
This is a phase III trial on Children. The investigators will enroll a total of 750 participants in Fajikunda Health Center (Gambia) The aims of the study are

* To describe the safety and immunogenicity of a booster dose of a licensed yellow fever vaccine administered to 3 different age cohorts of children, following a documented primary dose of a yellow fever vaccine administered at nine-months of age.
* To characterise the rate of yellow-fever PRNT sero-reversion (seropositive to seronegative) over a period of 9 months to 8 years following a single primary dose of yellow fever vaccine administered to Gambian infants at nine months age.
* To profile the immune response to the booster dose of YF vaccine in order to explore underlying mechanisms for longevity of vaccine-induced antibody.

DETAILED DESCRIPTION:
1. Background information and rationale

   1.2 Background information

   Yellow fever (YF) virus is a mosquito-borne flavivirus found in Sub-Saharan Africa and tropical South America. The virus causes YF, a viral haemorrhagic fever, which can be prevented by a highly effective live-attenuated vaccine, however, it is now considered a re-emerging disease due to the increased numbers of cases in the last 30 years.

   In most endemic countries across sub-Saharan Africa and South America, the YF vaccine is administered alongside other Expanded Programme on Immunization (EPI) vaccines, including the first measles containing vaccine (MCV1), at nine to 12 months of age. Several recent publications from Africa and Brazil have raised doubt that a single dose of YF vaccine will provide long lasting immunity: in a cohort vaccinated around nine-months of age in Ghana as part of a clinical trial of meningococcal vaccine, seropositivity, measured by microneutralization assay, had fallen from an already low 73%, 28 days following primary vaccination to 28% at 2.3 years . This figure had increased to 43% by six year - perhaps as a result of natural exposure or unrecorded re-vaccination. Our own data from samples collected in The Gambia and Mali 6 years post primary YF vaccinationadministered via the routine EPI program showed that 22.2% of a cohort of 467 children had undetectable antibody concentrations, with another 7.5% revealing concentrations below thethreshold of seropositivity of 0.5 IU/mL, confirming a substantial long-term decline in immunity relative to the early outcome of vaccination. Cross-sectional studies in Brazil, including nine month to 12-year olds, have similarly described a progressive decrease in the seropositivity rates from 87% within the first six-months after vaccination to 42% at six to eight years. It remains difficult to directly link the declining titres to actual occurrence of new cases of YF disease, as detailed immunisation history and in particular PRN titres are not available in observational studies of new cases, and no efficacy study has ever been performed. It is generally accepted though that high titres of YF antibodies protect against disease. The low residual titres in young children are therefore a legitimate cause for concern .

   1.2 Rationale Despite the vaccine being very successful at decreasing disease risk, YF is considered a re-emerging disease due to the increased numbers of cases in the last 30 years . Until 2014, the vaccine was recommended to be administered with boosters every 10 years, but in 2014 the World Health Organization recommended removal of booster doses for all except special populations . This recommendation has been questioned and there have been reports of waning antibody titers in adults over time and more recently also in paediatric populations. The scarcity of long-term studies on neutralising antibodies elicited in vaccinated infants has been identified as a knowledge gap in regard to the need for booster doses of the yellow fever vaccine. Based on these emerging data, the investigators need to establish whether infants who received a primary dose of a yellow fever vaccine at nine months of age, in line with EPI recommendations, are indeed likely to require a booster dose of the vaccine in order to ensure long-term protection.

   The investigators have a unique opportunity to address these questions of timing and immunogenicity which are of public health importance: The proposed trial leverages three well-characterized cohorts of infants in The Gambia, all of whom were vaccinated with the Institut Pasteur de Dakar 17D YF vaccine at nine to 10-months of age within. clinical trials run at the MRC Unit The Gambia at the London School of Hygiene and Tropical Medicine (MRCG). Details of the vaccine lots used and other metadata including anthropometric measurements and other health indices related to the infants at the time of vaccination are available. These trials are summarised in the table below and were all conducted with ethical approval at the MRC Unit in The Gambia and already have consent for future use of data and stored samples in the original ICDs.

   For most children in these cohorts, the initial serological responses to the vaccine are already documented from assays previously conducted at the Robert Koch Institute in Berlin, and for others serum samples from 28 days following the primary immunization remain in secure -80 storage. At the time of the study proposed, the cohorts will range in age from between 15 and 18 months, to between eight and nine years. These cohorts therefore provide a unique opportunity, not only to examine antibody decline over this time period, but also to determine the optimal timing of a booster dose following infant priming. In addition, they allow for comprehensive immune-profiling of innate and cellular responses to YF vaccination in the different age groups to generate new insights into determinants of long term immunity. Such data have never been generated in paediatric populations.

   1.3 Potential risks and benefits The risks are low as this is an already licensed vaccine and boosters have previously been recommended for adults with no safety concerns. The benefit is expected to be added protection against yellow fever infection based on an increase in PRNT titres, the established correlate of protection. Participants may also benefit from being assessed by a study clinician at the time of enrolment. Should any health complaints be identified during this screening initial treatment will be provided by the study team and the participant will be referred on for ongoing care, should this be necessary, at a government health facility.
2. Study objectives The main objective of this trial is to assess if a YF booster dose is required for children who received a single dose of YF vaccination in infancy and if so, at what age this booster dose might be most effective to administer.

   Primary • To describe the safety and immunogenicity of a booster dose of a licensed yellow fever vaccine administered to 3 different age cohorts of children, following a documented primary dose of a yellow fever vaccine administered at nine-months of age.

   Secondary
   * To characterise the rate of yellow-fever PRNT sero-reversion (seropositive to seronegative) over a period of 9 months to 8 years following a single primary dose of yellow fever vaccine administered to Gambian infants at nine months age.
   * To profile the immune response to the booster dose of YF vaccine in order to explore underlying mechanisms for longevity of vaccine-induced antibody.

   2.1 Study endpoints The primary endpoint of this study is the PRNT50 titres post booster vaccination according to intervals between primary YF vaccination and the booster dose.
3. Study design The proposed study leverages three well-characterized cohorts of infants, all of whom were vaccinated with the Institut Pasteur de Dakar 17D YF vaccine at nine to 10-months of age within clinical trials run within the Vaccines & Immunity Theme at the MRC Unit The Gambia at the London School of Hygiene and Tropical Medicine (MRCG) over the last few years.

   The databases of the previous trials, YF PRNT50 results from the primary immunisation and stored samples are immediately available to the investigators. Consent for sample storage and future work on remaining samples was obtained at the time of initial recruitment.

   3.1 Type of study and design This is a Phase 3 clinical trial to establish safety and immunogenicity of a booster dose of licensed YF vaccine in children of different age groups, following primary immunization with the same vaccine at 9-10 month of age.

   Children previously enrolled in each of the three historic vaccine trials (summarised in Table 1) will be recalled and invited for participation in the booster study. The investigators will enroll until 250 children will have been recruited per cohort. A roughly equal number of male and female participants will be enrolled in each cohort but no absolute percentage figures will be set.

   Following individual sensitization and informed consent, basic clinical and anthropometric data will be collected, and children will have a pre-booster blood sample (5.0-10 ml depending on age) obtained for YF PRNT50. All children will then receive a booster dose of the 17D YF vaccine manufactured by the Institut Pasteur de Dakar. All vaccines will be administered by the MRCG team. Local and systemic reactogenicity data will be solicited for 3 days. All children will then be invited back at day 28 (+7-day window) for a second blood sample (5.0-10 ml depending on age) and PBMC will be isolated and stored at the same timepoint. If, based on initial laboratory work, it is determined that a smaller number of PBMC will be required at this timepoint, only serum will be collected for post-booster YF PRNT50. A smaller cohort in each age group will be enrolled in the substudy described below.

   3.2 Sub-studies In order to conduct systems biology investigations which will provide novel insights into YF immune responses in children, subgroups of 30 children in each cohort will also be consented for a further sample (max. 5 ml) at either Day +7 for RNASeq or Day +14 for analysis of T cell responses - see below. The aim is to enrol the first 30 eligible children per cohort in the substudies, following consent provided on consent form version 1.0. Any child in these cohorts will have a maximum of 3 blood samples (up to 5 ml in the youngest age group, up to 10 ml/timepoint in the older age groups.)

   Humoral immune responses:

   Serum collected pre-and post YF vaccination will be separated from clotted whole blood samples, aliquoted and frozen at below -70°C prior to analysis at either the Institut Pasteur in Dakar or at the Robert Koch Institute in Berlin. This assay is not available in The Gambia. Post-primary serum from the primary studies is already available and safely stored for all participants and will also be analysed where data are not already available. Serum will be shipped using an IATA qualified shipping agent. A back-up sample will be retained at MRCG. Yellow Fever neutralizing antibody titres will be determined by a validated PRNT assay and results provided to MRCG for subsequent analysis.

   Cellular immune responses:

   To relate the serological responses to the B cell memory pool, Memory B cell Elispot assays will be carried out on fresh or banked PBMC from the V1 (baseline) and V2 (D+28 ) blood samples for all children where possible . PBMC will be isolated and stored. If, based on initial laboratory work, it is determined that a smaller number of PBMC will be required at this timepoint, serum will be collected alone.

   It is well established that both CD4 and CD8 T cell responses are elicited by YF vaccination, although their role in vaccine efficacy is not fully clarified. Recently published data in adults from a non-endemic setting have shown that both antibody and CD8 T cell responses might be impaired by a YF booster vaccine, compared to primary responses, however, there are no data in children.

   This study provides an excellent opportunity to further understand the impact of a booster dose on cellular immunity and its relationship-if any- to neutralising YF antibody. In addition to antibody analyses prior and post YF booster vaccination and saving of PBMC, subgroups of children (n=30) in each study cohort will therefore be sampled either at D+7 or D +14. On Day 7 whole blood samples (1-2 ml) will be collected into PaxGene tubes and analysed using RNASeq methodology, recently established in the Gambia. This method was recently applied to small volume blood samples of an infant cohort to understand immune ontogeny in unprecedented detail and will allow us to investigate whether YF antibody responses to the booster can be predicted by early "omic" signatures, as seen in adults. To date, this has not been studied in children. D+14 samples will serve to study cellular adaptive responses in via T cell profiling, ELISPOT assays and multi-parameter flow cytometry using established peptide pools and activation markers. T cell activation will be measured using the expression of CD69, CD38 and HLA-DR as well as the proliferation marker Ki67, in CD8 and CD4 T cells, using a protocol recently described . The determination of antigen-specific T cell responses via ELISPOT requires re-stimulation with peptide pools which the investigators will source commercially based on the published literature.

   All detailed "omic" and cellular immune studies can be implemented at the MRCG. Where possible, PBMC will be saved to test the hypothesis that the size of remaining B cell memory populations generated by primary YF immunisation will impact on the booster responses observed. The systems biology data generated will provide insights into the inter-relationship between early innate responses, T cell activation, B cell profiles and functional antibody. The investigators will use novel systems biology integrative approaches to inter-relate the immune-datasets, as recently published by the investigators. As has been shown by us and others, systems biology approaches not only permit the observation of a global picture of vaccine-induced innate immune responses but can also be used to predict the magnitude of the subsequent adaptive immune response and uncover new correlates of vaccine efficacy. This approach has not yet been applied to understanding YF immunity in children and is an exploratory element of the trial.

   3.3 Investigational products The vaccine to be used in this booster study is the licensed Institut Pasteur de Dakar 17D YF vaccine, which forms part of the National EPI program of The Gambia.

   3.3.1 Description of products This vaccine contains the Rockefeller17D-substrain 204 strain of Yellow fever virus. The exact potency of each batch is released with the certificate of analysis that accompanies each batch and the potency confirmed at time of release closest to internal minimum specification. This vaccine is the same vaccine used by the national EPI program.

   3.3.2 Formulation, packaging and labelling This vaccine is presented as a 10 dose vial with freeze-dried content which is reconstituted with a diluent, provided with the vaccine by the manufacturer.

   3.3.3 Product storage and stability The vaccine and diluent have to be kept at fridge temperature between +2/+8 degrees Celsius. The vaccine is supplied with a Vaccine Vial Monitor which will be used to determine wherther the vaccine is in a condition to be used at any point, including should any temperature deviations occur.

   3.3.4 Dosage, preparation and administration of investigational products Reconstituted vaccines have to be kept in a vaccine carrier at 2-8°C as per WHO and manufacturer requirements. Any remaining reconstituted vaccine not used has to be discarded after 6 h. The standard dose is 0·5 ml and is administered subcutaneously in the deltoid region using standard vaccination syringes (needle size 25G × 3/4") with a 45° injection angle.

   3.3.5 Concomitant medications/treatments Children due additional EPI vaccines during their period of enrolment in the study will have them administered following the day 28 blood sample. These vaccines will either be administered by the study team or the study team will ensure the vaccines are given through the routine EPI clinic at the site.

   No vaccines will be administered concomitantly with the yellow fever vaccines.
4. Selection and withdrawal of participants

   4.1 Selection of participants The study will recruit 750 healthy children to receive the booster dose of YF vaccine. Participants will be recruited/ re-approached from the previously enrolled participants in each of the vaccine trials.

   Upon screening, potentially eligible children will continue until end of study unless the trial is stopped for some reasons. A child may be excluded from the trial for the purposes of vaccination and/or clinical sampling or ongoing participation is considered to be against their best interests or if a contraindication to vaccination and/or to the obtaining of clinical samples is identified. Such decisions will be made by the PI in discussion with other members of the clinical trial team and/or sponsor. A child excluded in this way would be replaced and hence this would not alter the target sample size of 750. If not enough children from the previous cohorts are available, the investigators will aim to recruit appropriate age groups from community health centres. The investigators expect this to be an exception rather than the rule.

   4.2 Eligibility of participants Participants must meet all of the inclusion criteria and none of the exclusion criteria to be eligible to participate in the trial. A representative sample of children will be recruited from the target population.

   Potentially eligible children and their parents/guardian will be re-contacted

   4.2.1 Inclusion criteria Any child fitting the required age cohorts who has a documented record of having received a primary dose of the Institut Pasteur YF 17D vaccine between 9 and 12 months of age.

   Documented evidence can be either a previous record of YF vaccination with dates in our own trial registers if the child was a previous participant or documented evidence on the Infant Welfare card.

   4.2.2 Exclusion criteria • Any child with a height/length for weight z-score of -3 or below.

   • Any child known to be immunocompromised including any child with know vertical exposure to HIV infection.

   • Any child with a history of serious adverse event or other contraindication to previous yellow fever vaccination.

   • Participants who have an acute illness including abnormal vital signs or a fever of > 37.5°C will not be vaccinated on the day but may be invited back for rescreening when they have recovered.

   4.3 Withdrawal of participants

   A study participant will be discontinued from participation in the study if:
   * Any clinical significant adverse event (AE), intercurrent illness, or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the participant.
   * Development of any exclusion criteria.

   For further details on participant's premature termination see corresponding section below.

   Participants are free to withdraw from the study at any time without giving a reason.
5. Study procedures and evaluations

For an overview see the below"Schedule of Events". 5.1 Study schedule 5.1.1 Subject Identification and Sensitisation The databases of the previously conducted trials (summarized in table 1 above) will be accessed and interrogated for potentially available children according to age groups at the time of recruitment to the current booster study. Potentially suitable children according to the specified age cohorts will be identified and contact details for their families confirmed via Mobile phone calls. During such calls, it will be confirmed that the family is happy to be contacted for a further MRC study. If willingness to engage is confirmed, the broad details of the booster study are explained to the carer, and the carer and child will either be invited to a sensitization visit at the clinical trial site or via a home visit to share the informed consent document. The family is then given an appointment to attend the clinical trials site for Visit 1.

5.1.2 Enrollment Visit (Visit 1) At Visit 1, the Informed consent procedures will be completed and the eligibility criteria will be confirmed, vital signs and anthropomorphic data will be collected. The pre-booster blood sample will be collected and the booster dose of the YF vaccine administered as per protocol by the study team.

The child will be observed in the clinic for 30 minutes. At the end of 30 minutes it will be confirmed by a nurse to study clinician that the child remains well prior to them leaving clinic.

5.1.3 Follow-up Solicted adverse events (AE) will be collected up to and including Day 3 following the booster vaccination.

On Day 1, a member of the field team will conduct a home visit to assess and record any local or systemic AE including the presence of fever. Any child with a local or systemic response of concern will be reviewed by a study clinician the same day or within 24 hours according to the nature of the complaint. On Day 2 and 3 following vaccination, a member of the field team will contact the family by telephone to follow up on any ongoing or new local or systemic reaction. If there are any additional concerns, a home visit or clinic visit will be arranged as judged necessary by the study clinician. After Day 3 until end of study unsolicited adverse events will be collected. Parents will be asked to contact the study team and will be reviewed accordingly an safety data recorded.

Immunology subgroups:

Visit 1 +7 or 1 +14:

30 children per age cohort will be included in the immunology substudies which require a further blood sample on either Day 7 (+/-1) or Day 14 (+/-3) following the booster vaccination. To this purpose, the child will attend the clinic for blood sampling-see table below.

5.1.4 Final study visit On the final visit at Day 28 (+ 14 days), the child will be examined and a further blood sample of 5-10 ml will be collected (5 ml for children under 5 years old, up to 10 ml for older children).

5.2 Study evaluations

5.2.1 Clinical evaluations During Visit 1 and visit 2, clinical examination, vital signs, height and weight will be carried out and documented in the eCRF.

5.2.2 Laboratory evaluations No routine clinical laboratory blood samples will be collected in this study. The research blood samples will be collected on V1 and V2 for YF serology and B cell memory responses for which PBMC will be isolated and stored. If, based on initial laboratory work, it is determined that a smaller number of PBMC will be required at this timepoint, serum will be collected alone.

30 children per age cohort will be included in the immunology substudies which require a further blood sample on either Day 7 (+/-1) or Day 14 (+/-3) following the booster vaccination. To this purpose, the child will attend the clinic for blood sampling.

At any timepoint, a maximum of 5 ml of blood will be collected from children younger than 5 years of age, up to 10 ml from older children.

6 Safety considerations Yellow fever vaccines are generally exceptionally safe and have been given in millions of doses to adults and children worldwide. There have been rare reports of serious side-effects from the yellow fever vaccine. The rates for these severe 'adverse events following immunization' (AEFI), when the vaccine provokes an attack on the liver, the kidneys or on the nervous system are between 0 and 0.21 cases per 10 000 doses in regions where yellow fever is endemic, and from 0.09 to 0.4 cases per 10 000 doses in populations not exposed to the virus.

The risk of AEFI is higher for people with primary or secondary immune deficiency who will therefore be excluded from this study. In addition, any child with a history of serious adverse event to the previous yellow fever vaccine would be excluded from the booster study.

6.1 Methods and timing for assessing, recording, and analysing safety parameters

6.1.1 Adverse events An adverse event (AE) is any untoward medical occurrence in a study participant which does not necessarily have a causal relationship with either the vaccines administered or study participant. An AE therefore includes any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease occurring during the study period. Any AE which occurs after an immunization may be termed an AE following an immunization (AEFI).

For this trial, there will be active surveillance for local and/or systemic adverse events following immunization (AEFI) up to and including Day 3 following the booster vaccination. Established criteria will be used to record such events:

6.1.2 Reactogenicity Local solicited adverse event1 Based on the National Institute of Health, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events - Corrected Version 2.1 July 2017

6.1.3 Serious adverse events (SAEs)

An AE will be considered to be serious (I.e.. SAE) If:

* It results in death
* Is life-threatening1
* Requires in patient hospitalization or prolongations of existing hospitalization2.
* Results in persistent or significant disabilitiy

The start date for an SAE is defined as the day the relevant SAE criteria was met not the day an AE which subsequently developed into an SAE began. The end date for an SAE is the day the final AE resolves NOT the day the criteria rendering the AE serious resolves, i.e. if a articpant is admitted with dehydration secondary to gastroenteritis the SAE only ends when the diarrhoea resolves even if the infant has been discharged sometime before this. 'Death' and 'Persistent or significant disability/incapacity' will be defined as ongoing and will be closed for the purposes of further reporting once relevant clinical details have been captured (e.g. cause of death) and, in the case of disability/incapacity the condition is considered stable in the short term.

6.2 Reporting procedures SAE will be reported by the PI to the sponsor and the local safety monitor within 24 hours of the investigator team becoming aware. The report should be submitted on the designated SAE reporting form for the trial. The reports will be submitted by e-mail or via the online reporting form-dependign on MRCG SOP's. Follow-up reports will subsequently be submitted as new information becomes available until the SAE is closed or defined as ongoing.

Deaths occurring in the trial, irrespective of whether judged to be related or expected will be reported by the investigator by letter to the Gambia Government/MRCG joint ethics committee at their next meeting.

SAE that are judged to be related to investigational products and unexpected (SUSAR) will be reported by letter by the PI to The Gambia Government/MRCG Joint ethics committee within 24 hours.

SAE that are judged to be related to investigational products but not unexpected will be reported by letter by the PI to The Gambia Government/MRCG Joint ethics committee within 15 calendar days or within 7 calendar days if the event is fatal or life threatening.

All SAE will be reported by the PI to the Gambia Government/MRCG joint ethics committee in the annual report All deaths and all SAE that are judged to be related to investigational products will be reported to the Republic of the Gambia Medicines Control Agency by the sponsor according to the latest requirements of the agency.

If new information becomes available that may alter the safety or conduct of the trial the investigator will inform the sponsor, the Local Safety Monitor, The Gambia Government/MRCG Joint Ethics Committee and The Republic of the Gambia Medicines Control Agency in writing as soon as they become aware and generally within 5 calendar days.

6.3 Safety oversight This trial uses an already licensed product that is in general use in The Gambia with an established safety record. The product has also been used in booster vaccinations. The Trial is therefore considered as relatively low risk and given the background data and the short duration a DSMB is not judged to be required. A local safety monitor is in place nad will review local and systemic AE's and any SAE's, as will the trial management team on an ongoing basis.

7 Statistical considerations Sample size considerations

The primary endpoint of this study is the PRNT titres post booster vaccination according to intervals between primary YF vaccination and the booster dose. A sample size of 250 participants per cohort provides a precision of around + 5% over a range of plausible seroconversion rates associated with boosting at the three different timepoints (Table 2).

The same sample size also provides over 80% power to detect a 10% difference in the seroconversion/seroreversion rates between two different cohorts assuming a the rate in one of the cohorts compared of at least 85%. Also, over 90% power to detect a 15% difference in any two seroconversion/seroreversion rates.

Exploratory immunology studies:

Our previous systems biology studies showed that significant differences in "omic" signatures over the first week of life and according to day of life were detectable in cohorts of infants as small as n=10 per group. The investigators cannot currently confirm if such "omic" changes are informative to predict responses to YF vaccine in young children, but based on the data, systems biology approaches were informative in adults in group sizes as small as n=15. The investigators are therefore confident that a group size of 30 per sub-group will provide us with sufficient datasets to not only explore if "omic" signatures in children are also predictive of humoral responses to the booster, but also to interrogate pathways and cellular populations involved in mediating correlates of protection against yellow fever.

ELIGIBILITY:
Inclusion Criteria:

* Any child fitting the required age cohorts who has a documented record of having received a primary dose of the Institut Pasteur YF 17D vaccine between 9 and 12 months of age.
* Documented evidence can be either a previous record of YF vaccination with dates in our own trial registers if the child was a previous participant or documented evidence on the Infant Welfare card.

Exclusion Criteria:

* Any child with a height/length for weight z-score of -3 or below.
* Any child known to be immunocompromised including any child with know vertical exposure to HIV infection.
* Any child with a history of serious adverse event or other contraindication to previous yellow fever vaccination.
* Participants who have an acute illness including abnormal vital signs or a fever of > 37.5°C will not be vaccinated on the day but may be invited back for rescreening when they have recovered.

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Estimated)
Dates: Start 2022-05-16 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a PRNT (Plague Reduction Neutralization Testing) sero-conversion after receiving booster Yellow Fever vaccination. | 28 days post booster
  Children will receive Yellow fever booster vaccination and different intervals of the primary dose and their blood will be collected 28days after the booster and tested for seroconversion to PRNT.
Number of children who develop adverse events from Day 0 to D28 after receiving the booster Yellow fever vaccination | from Day 0 to Day 28 post booster
  After receiving the booster, children will be reviewed for adverse events 30 minutes to 1hour after the vaccination and followed up through home visits daily for 3days. Then they will be advised to come to the site for assessment if they develop an adverse event up to 28days after vaccination

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rezende IM, Sacchetto L, Munhoz de Mello E, Alves PA, Iani FCM, Adelino TER, Duarte MM, Cury ALF, Bernardes AFL, Santos TA, Pereira LS, Dutra MRT, Ramalho DB, de Thoisy B, Kroon EG, Trindade GS, Drumond BP. Persistence of Yellow fever virus outside the Amazon Basin, causing epidemics in Southeast Brazil, from 2016 to 2018. PLoS Negl Trop Dis. 2018 Jun 4;12(6):e0006538. doi: 10.1371/journal.pntd.0006538. eCollection 2018 Jun. PMID 29864115
- [Background] Domingo C, Fraissinet J, Ansah PO, Kelly C, Bhat N, Sow SO, Mejia JE. Long-term immunity against yellow fever in children vaccinated during infancy: a longitudinal cohort study. Lancet Infect Dis. 2019 Dec;19(12):1363-1370. doi: 10.1016/S1473-3099(19)30323-8. Epub 2019 Sep 19. PMID 31543249
- [Background] Idoko OT, Domingo C, Tapia MD, Sow SO, Geldmacher C, Saathoff E, Kampmann B. Serological Protection 5-6 Years Post Vaccination Against Yellow Fever in African Infants Vaccinated in Routine Programmes. Front Immunol. 2020 Oct 8;11:577751. doi: 10.3389/fimmu.2020.577751. eCollection 2020. PMID 33133096
- [Background] Campi-Azevedo AC, Reis LR, Peruhype-Magalhaes V, Coelho-Dos-Reis JG, Antonelli LR, Fonseca CT, Costa-Pereira C, Souza-Fagundes EM, da Costa-Rocha IA, Mambrini JVM, Lemos JAC, Ribeiro JGL, Caldas IR, Camacho LAB, Maia MLS, de Noronha TG, de Lima SMB, Simoes M, Freire MDS, Martins RM, Homma A, Tauil PL, Vasconcelos PFC, Romano APM, Domingues CM, Teixeira-Carvalho A, Martins-Filho OA. Short-Lived Immunity After 17DD Yellow Fever Single Dose Indicates That Booster Vaccination May Be Required to Guarantee Protective Immunity in Children. Front Immunol. 2019 Sep 26;10:2192. doi: 10.3389/fimmu.2019.02192. eCollection 2019. PMID 31616412
- [Background] de Noronha TG, de Lourdes de Sousa Maia M, Geraldo Leite Ribeiro J, Campos Lemos JA, Maria Barbosa de Lima S, Martins-Filho OA, Campi-Azevedo AC, da Silva Freire M, de Menezes Martins R, Bastos Camacho LA; Collaborative Group for Studies of Yellow Fever Vaccine. Duration of post-vaccination humoral immunity against yellow fever in children. Vaccine. 2019 Nov 15;37(48):7147-7154. doi: 10.1016/j.vaccine.2019.09.051. Epub 2019 Oct 4. PMID 31590934
- [Background] Vaccines and vaccination against yellow fever. WHO position paper -- June 2013. Wkly Epidemiol Rec. 2013 Jul 5;88(27):269-83. No abstract available. English, French. PMID 23909008
- [Background] Staples JE, Barrett ADT, Wilder-Smith A, Hombach J. Review of data and knowledge gaps regarding yellow fever vaccine-induced immunity and duration of protection. NPJ Vaccines. 2020 Jul 6;5(1):54. doi: 10.1038/s41541-020-0205-6. eCollection 2020. PMID 32655896
- [Background] Grobusch MP, Goorhuis A, Wieten RW, Verberk JD, Jonker EF, van Genderen PJ, Visser LG. Yellow fever revaccination guidelines change - a decision too feverish? Clin Microbiol Infect. 2013 Oct;19(10):885-6. doi: 10.1111/1469-0691.12332. Epub 2013 Aug 8. No abstract available. PMID 23927031
- [Background] Bovay A, Nassiri S, Maby-El Hajjami H, Marcos Mondejar P, Akondy RS, Ahmed R, Lawson B, Speiser DE, Fuertes Marraco SA. Minimal immune response to booster vaccination against Yellow Fever associated with pre-existing antibodies. Vaccine. 2020 Feb 24;38(9):2172-2182. doi: 10.1016/j.vaccine.2020.01.045. Epub 2020 Jan 31. PMID 32008879
- [Background] Kongsgaard M, Bassi MR, Rasmussen M, Skjodt K, Thybo S, Gabriel M, Hansen MB, Christensen JP, Thomsen AR, Buus S, Stryhn A. Adaptive immune responses to booster vaccination against yellow fever virus are much reduced compared to those after primary vaccination. Sci Rep. 2017 Apr 6;7(1):662. doi: 10.1038/s41598-017-00798-1. PMID 28386132
- [Background] Lee AH, Shannon CP, Amenyogbe N, Bennike TB, Diray-Arce J, Idoko OT, Gill EE, Ben-Othman R, Pomat WS, van Haren SD, Cao KL, Cox M, Darboe A, Falsafi R, Ferrari D, Harbeson DJ, He D, Bing C, Hinshaw SJ, Ndure J, Njie-Jobe J, Pettengill MA, Richmond PC, Ford R, Saleu G, Masiria G, Matlam JP, Kirarock W, Roberts E, Malek M, Sanchez-Schmitz G, Singh A, Angelidou A, Smolen KK; EPIC Consortium; Brinkman RR, Ozonoff A, Hancock REW, van den Biggelaar AHJ, Steen H, Tebbutt SJ, Kampmann B, Levy O, Kollmann TR. Dynamic molecular changes during the first week of human life follow a robust developmental trajectory. Nat Commun. 2019 Mar 12;10(1):1092. doi: 10.1038/s41467-019-08794-x. PMID 30862783
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Co MD, Terajima M, Cruz J, Ennis FA, Rothman AL. Human cytotoxic T lymphocyte responses to live attenuated 17D yellow fever vaccine: identification of HLA-B35-restricted CTL epitopes on nonstructural proteins NS1, NS2b, NS3, and the structural protein E. Virology. 2002 Feb 1;293(1):151-63. doi: 10.1006/viro.2001.1255. PMID 11853408
- [Derived] Kampmann B, Pley C, Strandmark J, Leigh MN, Ndow P, Clarke E, Roberts E, Faal A, Jeffries D, Kanteh E. Booster Vaccination against Yellow Fever in Gambian children-(BoVY) -a Phase 3 clinical trial to establish safety and immunogenicity of repeated YF vaccination in healthy Gambian children of different ages. Wellcome Open Res. 2024 Dec 24;9:733. doi: 10.12688/wellcomeopenres.23138.1. eCollection 2024. PMID 39935766